CLINICAL TRIAL: NCT00919776
Title: A Pilot Double Blind Controlled Study Randomizing Patients Whose ENL is Not Controlled With Standard Prednisolone, and Comparing a Group Treated With Ciclosporin to a Group Treated With Additional Steroid Only.
Brief Title: Ciclosporin in the Management of Chronic or Recurrent Erythema Nodosum Leprosum
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Homes and Hospitals of St Giles (Other); Alert Hospital, Ethiopia (Other); Armauer Hansen Research Institute, Ethiopia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITCCRBY24-ENLB
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Leprosy
Keywords: Leprosy; ENL; Erythema Nodosum Leprosum; Prednisolone; Ciclosporin
MeSH Terms: conditions — Leprosy | interventions — Prednisolone; Adrenal Cortex Hormones; Cyclosporine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ciclosporin (Experimental): ciclosporin reducing regimen lasting 16 weeks (additional prednisolone given for the first four weeks)
  Interventions: Drug: ciclosporin
- Prednisolone (Active Comparator): standard course of prednisolone given in a reducing regimen over 16 weeks
  Interventions: Drug: prednisolone

INTERVENTIONS:
Drug: prednisolone — prednisolone 40mg daily then reducing regimen over 16 weeks
  Other Names: corticosteroids
  Arms: Prednisolone
Drug: ciclosporin — Ciclosporin 7.5mg/kg - reducing regimen over 16 weeks (additional prednisolone given for the first four weeks)
  Other Names: Cyclosporine; Cyclosporin A
  Arms: ciclosporin

SUMMARY:
Study 2B: Ciclosporin in the management of chronic or recurrent Erythema Nodosum Leprosum Aim: To assess the safety, tolerability and efficacy of Ciclosporin in the treatment of patients whose ENL is not controlled with standard Prednisolone.

Objective: A pilot double blind controlled study randomizing patients whose ENL is not controlled with standard Prednisolone, and comparing a group treated with Ciclosporin to a group treated with additional steroid only.

DETAILED DESCRIPTION:
A pilot double blind controlled study randomizing patients whose ENL is not controlled with standard Prednisolone, and comparing a group treated with Ciclosporin to a group treated with additional steroid only.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with clinical evidence of recurrent or chronic ENL
* Aged 18-65
* Weigh more than 30Kg

Exclusion Criteria:

* Unwillingness to give informed consent
* Patients with severe active infections such as tuberculosis
* Pregnant or breastfeeding women (see Appendix II)
* Those with renal failure, abnormal renal function, hypertensive
* Patients taking thalidomide currently or within the last 3 months
* Patients not willing to return for follow-up
* Women of reproductive age not willing to use contraception for the duration of the study ( see Appendix II)
* HIV positive patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
number of ENL recurrence episodes per patient | up to 32 weeks

SECONDARY OUTCOMES:
Mean time to ENL recurrence after initial control | up to 32 weeks
Severity of ENL at recurrence | up to 32 weeks
Amount of additional prednisolone required by patients | up to 32 weeks
Frequency of adverse events for patients in each treatment arm | up to 32 weeks
Difference in score in Quality of Life assessment between start and end for patients in each treatment arm | up to 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Diana NJ Lockwood, MBChB, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Alert Hospital, Addis Ababa, Ethiopia